CLINICAL TRIAL: NCT04491604
Title: A Phase III Efficacy and Safety Study of Beremagene Geperpavec (B-VEC, Previously "KB103") for the Treatment of Dystrophic Epidermolysis Bullosa (DEB)
Brief Title: Ph 3 Efficacy and Safety of B-VEC for the Treatment of DEB
Acronym: GEM-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-VEC-03
Record Dates: First submitted 2020-07-22; First posted 2020-07-29 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-12

CONDITIONS: Dystrophic Epidermolysis Bullosa; Recessive Dystrophic Epidermolysis Bullosa; Dominant Dystrophic Epidermolysis Bullosa
Keywords: DEB
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Intervention Model Description: An intra-subject parallel study. Primary wounds are randomized within each subject, such that one wound receives B-VEC and the other wound receives placebo. Secondary wounds are selected to receive B-VEC only.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- B-VEC (Experimental): Topical gel of non-integrating, replication-incompetent HSV-1 expressing the human collagen VII protein
  Interventions: Biological: Topical Beremagene Geperpavec
- Placebo (Placebo Comparator): Matching masked inactive topical gel
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Topical Beremagene Geperpavec — Topical gel of non-integrating, replication-incompetent HSV-1 expressing the human collagen VII protein
  Arms: B-VEC
Other: Placebo — Matching masked inactive topical gel
  Arms: Placebo

SUMMARY:
To determine whether administration of topical B-VEC improves wound healing as compared to placebo, and to evaluate durability, repeat dosing (Primary Endpoint) and further obtain safety and tolerability data.

DETAILED DESCRIPTION:
Thirty-one (31) participants with DEB, aged 6 months or older at time of consent were enrolled for this Phase III study. The trial duration for each subject was about 6 months, with administration occurring once weekly. A Safety Follow-up Visit occurring 30 days from the date of final treatment with the Investigational Product also occurred. Each subject provided one pair of primary target wounds, with one wound from each pair randomized to be treated with B-VEC and the other wound with placebo. In addition to the primary target wound pair(s), additional wounds (secondary wounds) were selected to be treated with B-VEC. Throughout the study, participants complete questionnaires, had images captured of their study wounds, underwent physical exams, had vital signs and safety labs monitored.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or legally appointed and authorized representative must have read, understood and signed an Institutional Review Board/Ethics Committee (IRB/EC) approved Informed Consent or Assent Form and must be able to and willing to follow study procedures and instructions.
2. Age ≥ 6 months and older at the time of Informed Consent.
3. Clinical diagnosis of the Dystrophic Epidermolysis Bullosa.
4. Confirmation of DEB diagnosis (either DDEB or RDEB) by genetic testing including COL7A1.
5. Two (2) cutaneous wounds meeting the following criteria:

   1. Location: similar in size, located in similar anatomical regions, and have similar appearance
   2. Appearance: clean with adequate granulation tissue, excellent vascularization, and do not appear infected.
6. Subjects and caregivers who, in the opinion of the Investigator, are able to understand the study, co-operate with the study procedures and are willing to return to the clinic for all the required follow-up visits.
7. Male or Female of childbearing potential must use a reliable birth control method throughout the duration of the study and for three (3) months post last dose of B-VEC.
8. Negative pregnancy test at Visit 1 (Week 1), if applicable.

Exclusion Criteria:

1. Medical instability limiting ability to travel to the Investigative Center.
2. Diseases or conditions that could interfere with the assessment of safety and efficacy of the study treatment and compliance of the subject with study visits/procedures, as determined by the Investigator.
3. Current evidence or a history of squamous cell carcinoma in the area that will undergo treatment.
4. Subjects actively receiving chemotherapy or immunotherapy at Visit 1 (Week 1).
5. Active drug or alcohol addiction as determined by the Investigator.
6. Hypersensitivity to local anesthesia (lidocaine/prilocaine cream).
7. Participation in an interventional clinical trial within the past three (3) months (not including BVEC administration).
8. Receipt of a skin graft in the past three (3) months.
9. Pregnant or nursing women.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mission Dermatology Center, Rancho Santa Margarita, California
  - Stanford University, Stanford, California
  - Pediatric Skin Research, LLC, Coral Gables, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guide SV, Gonzalez ME, Bagci IS, Agostini B, Chen H, Feeney G, Steimer M, Kapadia B, Sridhar K, Quesada Sanchez L, Gonzalez F, Van Ligten M, Parry TJ, Chitra S, Kammerman LA, Krishnan S, Marinkovich MP. Trial of Beremagene Geperpavec (B-VEC) for Dystrophic Epidermolysis Bullosa. N Engl J Med. 2022 Dec 15;387(24):2211-2219. doi: 10.1056/NEJMoa2206663. PMID 36516090
- See also: Krystal Biotech, Inc. Patient and Family Advocacy Site — https://www.krystalbio.com/patients-and-families/patient-advocacy/

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Wounds
Groups:
- All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo"): Each subject provided one pair of primary target wounds, with one wound from each pair randomized to be treated with B-VEC and the other wound with placebo.
Period: Overall Study
Arm/Group | All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo")
Started | 31; 62 Wounds (Each subject provided one pair of primary target wounds, with one wound from each pair randomized to be treated with B-VEC and the other wound with placebo. The total primary wounds selected were 62 (=2x31), in which 31 each received B-VEC and Placebo, respectively. Additional wounds ("Secondary Wounds") were selected using the remaining weekly B-VEC dose. The number of Secondary Wounds treated depended on wound areas. The Secondary Wounds related data were not analyzed per protocol.)
B-VEC | 31; 31 Wounds
Placebo | 31; 31 Wounds
Completed | 28; 56 Wounds
Not Completed | 3; 6 Wounds
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo")
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.2 (10.70)
Age, Customized [Count of Participants; unit: Participants]
  <= 12 years | 10
  > 12 and <= 18 years | 9
  > 18 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31
Primary Wound Area(cm^2) B-VEC [Mean (Standard Deviation); unit: cm^2] | 14.354 (12.6930)
Primary Wound Area(cm^2) Placebo [Mean (Standard Deviation); unit: cm^2] | 15.565 (12.1315)

OUTCOME MEASURES:

1. Primary Outcome: Primary Wound With Complete Wound Healing (100% Wound Closure) on Weeks 22 and 24 or Weeks 24 and 26
Description: The primary wound was defined as a responder wound that met either of the following conditions:
  * Complete wound healing on Week 22 and Week 24, or
  * Complete wound healing on Week 24 and Week 26.
  For subjects with missing primary wound healing data, a multiple imputation approach (10 repliates) was used. The total numbers of primary wounds with complete healing for B-VEC and Placebo presented below were the average of those from the multiple imputation replicates, and therefore, they would not be whole numbers (integers).
Time Frame: 26 weeks post-baseline
Population: The intent-to-treat (ITT) population included subjects whose primary wounds were randomized regardless of whether they received randomized treatment or not.
Measure: Number; unit: number of wounds with complete healing
Units Other Than Participants: Wounds
Arm/Group | B-VEC | Placebo
Number analyzed (Participants) | 31 | 31
Number analyzed (Wounds) | 31 | 31
number of wounds with complete healing | 20.9 | 6.7
Statistical Analysis 1: Comparison: B-VEC vs Placebo; The null hypothesis of interest was the absence of a treatment effect on wound healing and the alternative hypothesis is the presence of a treatment effect on wound healing. The Hypothesis was tested by exact McNemar's test on the paired primary wound healing data. For subjects with missing primary wound healing data, a multiple imputation approach was used; Test type: Equivalence — The Hypothesis was tested by exact McNemar's test on the paired primary wound healing data; p = 0.00192, McNemar; The Hypothesis was tested by exact McNemar's test on the paired primary wound healing data. A multiple imputation approach was used for missing data; responder rate difference = 45.8, 95% CI 2-sided [23.6 to 68.0] — The difference is the treatment/discordance difference in percentage of responders (primary wounds with complete healing), which is the same as the difference in the percentage of treatment responders and the percentage of placebo responders

2. Secondary Outcome: Primary Wound With Complete Wound Healing (100% Wound Closure) on Weeks 8 and 10 or Weeks 10 and 12
Description: The primary wound was defined as a responder wound that met either of the following conditions:
  * Complete wound healing on Week 8 and Week 10, or
  * Complete wound healing on Week 10 and Week 12.
  For subjects with missing primary wound healing data, a multiple imputation approach (10 repliates) was used. The total numbers of primary wounds with complete healing for B-VEC and Placebo presented below were the average of those from the multiple imputation replicates, and therefore, they would not be whole numbers (integers).
Time Frame: 12 weeks post-baseline
Population: as for outcome 1
Measure: Number; unit: number of wounds with complete healing
Units Other Than Participants: Wounds
Arm/Group | B-VEC | Placebo
Number analyzed (Participants) | 31 | 31
Number analyzed (Wounds) | 31 | 31
number of wounds with complete healing | 21.9 | 6.1
Statistical Analysis 1: Comparison: B-VEC vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The Hypothesis was tested by exact McNemar's test on the paired primary wound healing data; p = 0.00047, McNemar — There is no multiplicity adjustment needed since the hypothesis testing are hierarchical; [statistical method as in outcome 1, analysis 1]; responder rate difference = 51.0, 95% CI 2-sided [29.3 to 72.6] — The difference is the treatment/discordance difference in percentage of responders (complete wound healing), which is the same as the difference in the percentage of treatment responders and the percentage of placebo responders

3. Secondary Outcome: Primary Wound Pain Severity (Visual Analog Scale (VAS)) Change for Ages 6 and Above Subjects at Weeks 22, 24, and 26.
Description: Changes from baseline at Weeks 22, 24, and 26 in primary wound pain severity (visual analog scale (VAS)) for ages 6 and above subjects. The Visual Analog Scale scores from 0 (no pain) to 10 (the worst possible pain). Negative values in changes from baseline mean improvement in pain severity.
Time Frame: 26 weeks post-baseline
Population: The intent-to-treat (ITT) population included subjects whose primary wounds were randomized regardless of whether they received randomized treatment or not. For pain severity, only subjects ages 6 and above were evaluated (n=27). The analyses were based on observed data where missing data were not imputed, therefore the numbers of available data for analyses could be less than the total.
Measure: Mean (Standard Deviation); unit: score on a scale of 0 to 10
Arm/Group | B-VEC | Placebo
Number analyzed (Participants) | 27 | 27
score on a scale of 0 to 10
  Week 22: number analyzed (Participants) | 24 | 24
  Week 22 | -0.88 (2.346) | -0.71 (2.476)
  Week 24: number analyzed (Participants) | 25 | 25
  Week 24 | -0.64 (2.325) | -0.08 (2.548)
  Week 26: number analyzed (Participants) | 24 | 24
  Week 26 | -0.63 (2.123) | -0.38 (2.871)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo"): Each subject provided one pair of primary target wounds, with one wound from each pair randomized to be treated with B-VEC and the other wound with placebo. Due to the 'split-person'/intrasubject design, each subject received both B-VEC and Placebo. Therefore, the safety assessments were reported at subject level, but not per intervention.
Arm/Group | All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo")
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 3/31
Other Adverse Events (participants affected / at risk) | 17/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo") (N=31)
Cellulitis (Infections and infestations) | 1 (1) — cellulitis of the right leg
Diarrhoea (Gastrointestinal disorders) | 1 (1) — Diarrhoea
Anaemia (Blood and lymphatic system disorders) | 1 (2) — severe anemia
Blood culture positive (Investigations) | 1 (1) — Blood culture positive
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo") (N=31)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Chills (General disorders) | 3 (3)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT04491604/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT04491604/SAP_001.pdf